CLINICAL TRIAL: NCT00470301
Title: A Phase I-II Study of R115777 (Tipifarnib, Zarnestra®) Plus Sequential Weekly Paclitaxel Followed by Dose-Dense Doxorubicin and Cyclophosphamide in Patients With Stage IIB-IIIC Breast Cancer
Brief Title: Tipifarnib and Combination Chemotherapy in Treating Patients With Stage II or Stage III Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00239; NCI-2009-00239 (Other: CTRP (Clinical Trial Reporting Program)); 06-12-487 (Other: Montefiore Medical Center); 7868 (Other: CTEP); P30CA013330 (NIH); N01CM62202 (NIH); N01CM62204 (NIH)
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Male Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — tipifarnib; Paclitaxel; Taxes; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Tipifarnib plus sequential weekly paclitaxel followed by doxorubicin plus cyclophosphamide
  Interventions: Drug: tipifarnib; Drug: paclitaxel; Drug: doxorubicin; Drug: cyclophosphamide

INTERVENTIONS:
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: doxorubicin — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana

SUMMARY:
Tipifarnib may stop the growth of breast cancer by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as paclitaxel, doxorubicin, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving tipifarnib together with combination chemotherapy may kill more tumor cells. This phase I/II trial is studying the side effects and best dose of tipifarnib when given together with combination chemotherapy and to see how well they work in treating patients with stage II or stage III breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose of tipifarnib when given together with paclitaxel in patients with stage IIB-IIIC breast cancer. (Phase I) II. To determine the pathologic complete remission rate (including breast and breast plus axillary nodes) in patients treated with sequential paclitaxel and tipifarnib followed by dose-dense doxorubicin hydrochloride, cyclophosphamide, and tipifarnib. (Phase II) III. To determine the feasibility and safety of this regimen in these patients. (Phase I and II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of tipifarnib followed by a phase II study.

PHASE I: Paclitaxel plus tipifarnib: Patients receive paclitaxel IV over 1 hour on day 1 and oral tipifarnib twice daily on days 1-3.

Treatment repeats weekly for 12 courses in the absence of disease progression or unacceptable toxicity. Patients with no evidence of disease progression after 12 courses proceed to AC chemotherapy plus tipifarnib. Cohorts of 3-6 patients receive escalating doses of tipifarnib until the recommended phase II dose (RTPD) is determined. The RTPD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

AC chemotherapy plus tipifarnib: Patients receive doxorubicin hydrochloride IV over 5-10 minutes and cyclophosphamide IV over 30-60 minutes on day 1, oral tipifarnib twice daily on days 2-7, and pegfilgrastim subcutaneously on day 2.

Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients receive paclitaxel and tipifarnib at the RTPD and AC chemotherapy plus tipifarnib as in phase I. After completion of AC plus tipifarnib (in both phases), patients are re-evaluated for surgery (i.e., modified radical mastectomy, radical mastectomy, segmental mastectomy or lumpectomy with an axillary lymph node dissection).

After completion of study treatment, patients are followed every 6 months for 5 years and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast; clinical stage IIB, IIIA, IIIB, or IIIC disease
* At least 1 week since prior tamoxifen or other selective estrogen receptor modulator for prevention or for other indications (e.g., osteoporosis or prior ductal carcinoma in situ)
* HER-2/neu-negative by immunohistochemistry or fluorescence in situ hybridization (FISH)
* Hormone receptor status:

  * Estrogen and/or progesterone receptor-positive* [Note: *Patients enrolled on the phase I portion of the trial may have estrogen and progesterone receptor-negative disease]
* Normal organ function including:
* WBC >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin normal
* AST and ALT =< 2.5 times upper limit of normal
* LVEF normal by echocardiogram or nuclear scan
* Creatinine normal OR Creatinine clearance >= 60 mL/min
* FEV1 >= 1 L* and DLCO >= 50%* [Note: *Only if baseline CT scan of chest shows parenchymal lung disease OR there is a history of chronic obstructive or other pulmonary disease]
* No prior chemotherapy, radiotherapy, or definitive therapeutic surgery (e.g., mastectomy, lumpectomy, or axillary dissection) for this cancer but prior sentinel lymph node biopsy for this malignancy allowed
* No prior adjuvant chemotherapy for a previous breast malignancy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* ECOG performance status 0-1
* Fertile patients must use effective contraception

Exclusion criteria:

* No other invasive malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to tipifarnib or other study drugs (e.g., imidazoles or quinolones)
* No other uncontrolled illness including, but not limited to, any of the following: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would preclude study compliance
* Not pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, Principal Investigator — Montefiore Medical Center
Locations (7):
- United States (7):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Andreopoulou E, Vigoda IS, Valero V, Hershman DL, Raptis G, Vahdat LT, Han HS, Wright JJ, Pellegrino CM, Cristofanilli M, Alvarez RH, Fehn K, Fineberg S, Sparano JA. Phase I-II study of the farnesyl transferase inhibitor tipifarnib plus sequential weekly paclitaxel and doxorubicin-cyclophosphamide in HER2/neu-negative inflammatory carcinoma and non-inflammatory estrogen receptor-positive breast carcinoma. Breast Cancer Res Treat. 2013 Oct;141(3):429-35. doi: 10.1007/s10549-013-2704-x. Epub 2013 Sep 26. PMID 24068539

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: See Detailed Description
  tipifarnib: Given orally
  paclitaxel: Given IV
  doxorubicin hydrochloride: Given IV
  cyclophosphamide: Given IV
  pegfilgrastim: Given SC
  conventional surgery: surgical procedures performed on patients
  axillary lymph node dissection: correlative study
Period: Overall Study
Arm/Group | Arm I
Started | 60
Completed | 55
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate (pCR)
Description: An increase in the breast pCR from 15% (anticipated for chemotherapy alone) to 35% would be considered promising.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 55
participants | 33 [7 to 36]

2. Primary Outcome: Number of Participants Analyzed for Phase II Dose of Tipifarnib When Combined With Weekly Sequential Paclitaxel (Phase I)
Description: The recommended phase II dose of tipifarnib (100 or 200 mg PO BID on days 1-3 each paclitaxel dose) in combination with paclitaxel (80 mg/m2/week x 12 consecutive weeks)
Time Frame: 1 year
Population: Total participants analyzed is 6. 3 received 100 mg PO BID tipifarnib and 3 received 200 mg PO BID tipifarnib.
Measure: Number; unit: participants
Arm/Group | Arm I
Number analyzed (Participants) | 6
participants
  Number of participants with DLT (100 mg PO BID tipifarnib): number analyzed (Participants) | 3
  Number of participants with DLT (100 mg PO BID tipifarnib) | 0
  Number of participants with DLT (200 mg PO BID tifiparnib): number analyzed (Participants) | 3
  Number of participants with DLT (200 mg PO BID tifiparnib) | 0

ADVERSE EVENTS:
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 13/60
Other Adverse Events (participants affected / at risk) | 28/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=60)
Neutropenia (Blood and lymphatic system disorders) | 13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=60)
Fatigue (General disorders) | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less